CLINICAL TRIAL: NCT03392090
Title: SHARE (Sharing Goals and Preferences) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Nancy L. Keating, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-520
Record Dates: First submitted 2017-12-20; First posted 2018-01-05 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Other Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- More Good Days video&brief questionnaire (Experimental): * Participants will watch the More Good Days video and will be given a brief questionnaire and wallet card to help identify their goals and preferences about information and care
  * The More Good Days video is developed to help patients with advanced cancer think about what a good day means to them and to help them think about questions they may have for their physicians when discussing treatments.
  * The 3-page brief questionnaire is designed to help patients identify their preferences about information and care and to help encourage a conversation between patients and their doctors and health care team about their goals and preferences
  * The wallet card will help patients think about questions they may want to ask their providers when considering treatments.
  Interventions: Other: More Good Days video&brief questionnaire

INTERVENTIONS:
Other: More Good Days video&brief questionnaire — Help patients with advanced cancer think about what a good day means to them and to help them think about questions they may have for their physicians when discussing treatments

SUMMARY:
This research study is evaluating the usefulness of a video and questionnaire to help cancer patients think about the goals of their care.

DETAILED DESCRIPTION:
The investigators are conducting a study with patients from Dana Farber Cancer Institute (DFCI) and DFCI-affiliate at St. Elizabeth's Hospital who are being treated for their cancer. The purpose of the study is to test the implementation of a short video, a brief questionnaire, and a wallet card designed to help patients understand and articulate their goals and preferences when making decisions about their cancer treatment and communicate these preferences to their clinicians.

The short video and brief questionnaire were developed to help patients with cancer think about their goals of care and their treatment and information preferences and to prompt discussions with their health care team about these preferences. The wallet card is designed to help patients remember some key questions that may be useful as they make decisions about future treatments

A pilot test will be completed to assess the feasibility and usability of the revised "More Good Days" video, brief questionnaire and wallet card in helping seriously-ill cancer patients think about what a good day means to them and test whether these tools can help patients to identify and communicate their medical treatment preferences and goals with their care team.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are receiving treatment at:

  * DFCI in the thoracic oncology group
  * DFCI-affiliated St. Elizabeth's Hospital and have progressed on 2nd line or later-line systemic therapies (chemotherapy, immunotherapy, biological, or targeted therapies)
* Clinicians' schedules to identify patients with metastatic cancers who are considering or pursuing additional palliative therapy

Exclusion Criteria:

* Patients who are not interested in the study
* Patients of physicians who opt out of participating
* Patients whose physicians did not opt out, but whose physician does not think they are well suited for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Enrollment | 2 years
  % of patients invited to participate who choose to enroll
Overall rating of intervention | 1 month
  % who rate intervention as good/very good/excellent.
Would recommend intervention to others | 1 month
  % who would recommend intervention to others with cancers like theirs

SECONDARY OUTCOMES:
Preferred format for viewing video and completing questionnaire | 1 month
  preferences for watching alone vs. with family; in clinic vs. home, interest in accessing via electronic record portal
Patient anxiety | 1 month
  Hospital Anxiety and Depression Scale (HADS) (score 0 to 21 for 7 anxiety items, higher=more anxiety)
Patient distress | 1 month
  National Comprehensive Cancer Network distress thermometer (score 0 to 10, higher worse distress)
Patient depression | 1 month
  Patient Health Questionnaire-9 (PHQ-9) (9 items, score 0 to 27, higher = more depressed)
Hope | 1 month
  Hearth Hope Index (12 items, score 12 to 48, higher = more hope)
FACIT-PAL Quality of Life | 1 month
  FACIT-PAL instrument general quality of life (27 general items, score 0 to 108, higher=better quality of life)
Quality of life-palliative care specific items | 1 month
  Palliative care subscale of FACITPAL (14 items, score 0 to 56, higher = better quality of life)
Therapeutic Alliance | 1 month
  Human Connection Scale (16 items, score 16 to 64, higher = more therapeutic alliance)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Keating, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute at St Elizabeth, Boston, Massachusetts
  - Nancy Keating, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wright AA, Thompson E, Nguyen MV, Wescott P, Barry MJ, Lathan CS, Keating NL. The SHARE Study: Pilot Study of a Communication Intervention Designed to Elicit Advanced-Stage Cancer Patients' Preferences and Goals. J Palliat Med. 2022 Nov;25(11):1646-1654. doi: 10.1089/jpm.2021.0655. Epub 2022 Jun 23. PMID 35736783